CLINICAL TRIAL: NCT06807476
Title: Turkish Validity and Reliability of the Acupuncture Readiness Attitude Scale
Brief Title: Turkish of the Acupuncture Readiness Attitude Scale
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Collaborators: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Head of Department of Obstetrics and Gynecology Nursing, Bartın Unıversity
Other Study IDs: 2024-SBB-0605
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Acupuncture; Reliability and Validity
Keywords: Turkish
MeSH Terms: interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validity and reliability
  Interventions: Other: Validity and reliability

INTERVENTIONS:
Other: Validity and reliability — The scale consists of 40 items and four sub-dimensions, and is scored according to a 5-point Likert rating scale (ranging from "Strongly Disagree" (Score = 1 point) to "Strongly Agree" (Score = 5 points)). The scale evaluates the healthy/patient individual's readiness attitude level towards acupuncture, personal beliefs, preferences and experiences. The score received per sub-dimension varies between a minimum of 10 and a maximum of 50 points. The average cut-off score per sub-dimension is 25. The higher the score (above the average cut-off score), the more open the healthy/patient individual is to acupuncture. Sub-dimensions:
  Sub-Dimension 1 (Items 1-10): Willingness to Try Acupuncture Sub-Dimension 2 (Items 11-20): Belief in the Effectiveness of Acupuncture Sub-Dimension 3 (Items 21-30): Comfort in the Acupuncture Sub-Dimension 4 (Items 31-40): Concerns and Preferences

SUMMARY:
Objectives: Acupuncture is often used to promote health and well-being, relieve pain, and treat a variety of medical conditions. Acupuncture is believed to work by stimulating the body's natural healing processes, and it is important that individuals are prepared to receive acupuncture. The study aims to examine the Turkish validity and reliability of the Acupuncture Readiness Attitude Scale, which will be used to evaluate the well-being levels of haptonomy and haptotherapy practices in women.

Design: The study was methodological type. Methods: The study conducted between Aug 9 and December 30, 2024, with 510 women who volunteered to participate by sharing forum pages on social media (Facebook, Instagram) via the web. Data were collected using a personal information form, including sociodemographic and obstetric characteristics and the Acupuncture Readiness Attitude Scale.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are over the age of 18,
* Live in Turkey,
* Use social media, and agree to participate in the study will be included in the study.

Exclusion Criteria:

* Women who do not know how to read or write Turkish,
* Have hearing or vision problems or mental disabilities,
* Do not have social media,
* Do not volunteer to participate in the study will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women over 18 age, living in Turkiye, using social media (Facebook, Instagram), and agreeing to participate in the study
Sampling Method: Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The Acupuncture Readiness Attitude Scale | 1 day
  The scale consists of 40 items and four sub-dimensions, and is scored according to a 5-point Likert rating scale (ranging from "Strongly Disagree" (Score = 1 point) to "Strongly Agree" (Score = 5 points)). The scale evaluates the healthy/patient individual's readiness attitude level towards acupuncture, personal beliefs, preferences and experiences. The score received per sub-dimension varies between a minimum of 10 and a maximum of 50 points. The average cut-off score per sub-dimension is 25. The higher the score (above the average cut-off score), the more open the healthy/patient individual is to acupuncture.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No